CLINICAL TRIAL: NCT02585882
Title: Caries Preventive Effect of Salt Fluoridation in Preschool Children in The Gambia
Brief Title: Preventive Effect of Salt Fluoridation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, PD Dr. A. Rainer Jordan, Priv.-Doz. Dr. med. dent. habil., MSc., University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1062010
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Fluorides, Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Communal preschool feeding with fluoridated salt (Experimental): According to the allocation concealment, subjects of the test group were preschool children at the "Kindergarten Wattenscheid in Gambia", Brikama-Kabafita, West Coast Region, The Gambia.
  Interventions: Other: Fluoride table salt
- Communal preschool feeding with no fluoridated salt (No Intervention): Subjects of the control group were preschool children at the "Kindergarten Bottrop in Gambia", Brikama, West Coast Region, The Gambia.

INTERVENTIONS:
Other: Fluoride table salt
  Arms: Communal preschool feeding with fluoridated salt

SUMMARY:
This was a block-randomized, controlled, open-label trial and was executed in two preschools in The Gambia. Fluoridated table salt (250 mg F/kg salt) was administered in daily communal preschool feeding. In total, 304 children in the test group and 137 children in the control group, aged 3 to 5 years were enrolled according to inclusion criteria (complete primary dentition and a parental or legal guardian informed consent). Mean difference of incidence of cavitated carious lesions (Δd3/4mft) after 12 months was the primary end point. The relative preventive dental caries effect was. Secondary end points were the difference of incidence of white spot lesions and the difference of incidence of total carious lesions.

DETAILED DESCRIPTION:
Patients and Methods This was a block-randomized, controlled, open-label trial to evaluate the relative caries preventive effect of fluoridated table salt in communal feeding of preschool children after 12 months. The study protocol was approved by the Witten/Herdecke University institutional review board (No. 106/2010) and by the Department of State for Health and Social Welfare of the Republic of The Gambia in the form of a memorandum of understanding. All participants and parents or legal guardians gave written informed consent with the aid of a native speaker before study-related procedures were performed and the study was conducted in line with the Declaration of Helsinki. Figure 1 describes the study design in brief.

Sample Size Sample size calculation was performed with G*Power 3. Basic data for sample size calculation was the mean dental caries experience of preschool children in urban parts of The Gambia that was reported to be 2.09 dmft teeth (SD: 1.92). An effect measure of caries prevention by fluoridated table salt of 35 % was assumed according to the relevant literature. Alpha error was set with 0.05, and the study power with 80 %. A target sample of 130 subjects for each study arm (test and control group) was calculated.

Study Population

Eligible participants were children aged from 3 - 5 years living in urban Gambia with preschool attendance at the co-operating kindergartens. The inclusion criteria for participating in this study were:

1. a complete primary dentition
2. parental or legal guardian informed consent. The only exclusion criteria was refusal to participate in the study. Study End Points To measure the caries preventive effect of salt fluoridation (1) the difference of incidence of cavitated carious lesions (Δd3/4mft) after study related intervention was chosen as the primary end point. Using the primary study end point, the relative preventive dental caries effect was calculated according to the following formula: 100 - (Δd3/4mft (test group) / Δd3/4mft (control group)) x 100.

Secondary end points were:

(2) the difference of incidence of white spot lesions (ΔG2-4) with G2 denoting slight white spot formation, G3 denoting excessive white spot formation, and G4 denoting white spot formation with cavitation into enamel.

(3) the difference of incidence of total carious lesions (ΔTCL (= G2-4 + d3/4mft)).

Total carious lesions (TCL) were calculated as a weighted sum score according to the following weights: G2: 1 point; G3: 2 points; G4: 3 points; d3/4t and ft: 4 points; tooth with pulpitis, ulcera, fistula or abscess due to caries: 5 points; missing tooth (mt): 6 points.

For quality control, (4) a fluoride concentration measurement of the table salt was performed as safety endpoint at t0, t0+6 mths, and t0+12 mths = t1. For this purpose, packages with fluoridated salt and provided for the study were randomly selected. Measurements were executed using an Orion Ionplus Fluoride Electrode (Thermo Electron, Beverly, USA) after standardised calibration for low-level measurement. The analysis was undertaken in triplicate per sample, and a mean was calculated for each measurement point. The threshold limit value was set at 0.1 ppm F-.

Participants and Investigators Participants were screened, recruited, and included in the study at two public preschools in Brikama, West Coast Region, The Gambia, in March 2012. The screening and dental examinations took place during regular teaching time in an affiliated dental station. Two investigation teams performed the study related examinations. A team consisted of two dentists of which one was the clinical investigator and the other served as information specialist. All were equally calibrated in clinical dental caries screening. Inter-examiner Cohen´s reliability Ҡ was 0.82 [Cohen, 1960], indicating an almost perfect match against the expert (RAJ).

Randomization and Allocation Concealment As the intervention procedure was bound to the communal preschool feeding, an individual randomization of subjects to the study arms was not feasible. Instead, one preschool was chosen for intervention and the other preschool served as control. The assortment of intervention was performed according to a random selection by a person who apart from this was not involved in the study (LGW). All preschool children meeting inclusion and exclusion criteria were primarily allocated to the test group and to the control group, respectively.

Interventions Natural fluoride availability in the Gambian West Coast Region had been determined in advance of this interventional study to evaluate general fluoride availability. In the study region, the fluoride concentration in drinking water was determined to be 0.1 mg/liter. In this region, traditional oral hygiene for children does not comprise (fluoride) toothpastes until religious maturity at the age of about 12 years.

Study related intervention of administration of fluoridated table salt (MarkenJodSalz + Fluorid, Südsalz, Heilbronn, Germany) was organised during once-daily communal preschool feeding. Acccording to the manufacturer's declaration, fluoride concentration of the fluoridated table salt was 250 mg/kg. The central preschool kitchen was instructed to flavour the meals with a calculated amount of fluoridated table salt. The amount was set with 0.4 mg fluoride per capita and day for a period of 12 months. The study intervention period was executed between September 2012 and August 2013. The calculation for the total flavouring table salt amount was as follows:

* number of subjects in the intervention preschool (including subjects not included in the study but taking part in the communal preschool feeding) n = 450
* fluoride concentration of fluoridated table salt: 25 mg F- per 100 g salt
* recommended daily age-dependent supplementary dose: 0.4 mg fluoride per capita (i. e. 0.05 - 0.07 mg F- per kg body weight)
* consequently, 720 g fluoridated table salt daily for preparation of the communal preschool feeding, resp. 1.6 g fluoridated table salt per capita and day, which complied with recent WHO recommendations of salt intake.

Meals of the control group were prepared without fluoridated table salt. Before starting the intervention, all subjects received a dental examination at t0. Teeth were cleaned with an electric toothbrush (Vitality precision clean, Oral-B, Schwalbach, Germany) before inspection without using toothpaste. Teeth were then dried with cotton rolls (Cotton rolls for kids, Roeko, Langenau, Germany) and hand-bellows (Delamax, Berlin, Germany). Dental caries inspection was performed visually with the aid of dental mirrors and blunt probes in natural light according to recent recommendation for epidemiological field studies. With respect to available field hygiene measures, disposable dental instruments were used (Nordenta, Hamburg, Germany). After completion of the intervention, all subjects were dentally examined again at t1 in the exact same manner than at t0.

Study Settings According to the allocation concealment, subjects of the test group were preschool children at the "Kindergarten Wattenscheid in Gambia", Brikama-Kabafita, West Coast Region, The Gambia. Subjects of the control group were preschool children at the "Kindergarten Bottrop in Gambia", Brikama, West Coast Region, The Gambia.

Study Hypothesis The investigators used a null hypothesis (H0) assuming no statistical difference of Δd3/4mft at t1 between the test group and control group.

Statistical Analysis Demographic data were compared as inter group comparison using Wilcoxon rank sum test with p <0.05 for statistical significance. Analyses of the study end points were performed using 95 percent confidence intervals (95%-CI). IBM SPSS software (version 21; International Business Machines Corp, Armonk, USA) was used for computing statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. a complete primary dentition
2. parental or legal guardian informed consent.

Exclusion Criteria:

* refusal to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
caries increment | 12 months
  difference of incidence of cavitated carious lesions (Δd3/4mft)